CLINICAL TRIAL: NCT07350109
Title: An Explorative Prospective Non-interventional Study on Sedation Depth in Postoperative Cardiac Surgery Patients Using Blinded BIS Monitoring
Brief Title: Investigation of Sedation Depth Via BIS Monitoring in ICU After Cardiac Surgery
Acronym: BISICU
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 1368
Record Dates: First submitted 2025-11-24; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Sedation After Cardiac Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: adult patients who have undergone cardiac surgery expected to require invasive mechanical ventilation and continuous sedation for more than six hours postoperatively

SUMMARY:
This study is a non-interventional, observational research project focused on monitoring sedation levels in patients who have undergone cardiac surgery. It uses a tool called Bispectral Index (BIS), which measures brain activity to assess sedation depth. The goal is to understand how often patients experience deep sedation (BIS <50) during the first 48 hours in the ICU and to explore its impact on clinical outcomes like ventilation duration, ICU stay length, and complications such as infections or delirium.

The study is conducted at two hospitals in Austria and involves patients who require mechanical ventilation and continuous sedation for more than six hours after surgery. BIS data will be collected continuously, but the readings will be blinded to the clinical team, meaning they will not influence patient care. Sedation will be managed using standard clinical practices.

The findings aim to improve sedation management in ICUs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Undergoing cardiac surgery with subsequent admission to the ICU
* expected duration of invasive mechanical ventilation > 6 hours postop.
* Written informed consent obtained from the patient or legal representative (if the patient is not capable of consent).

Exclusion Criteria:

* Pre-existing neurological disorders affecting consciousness or sedation assessment (e.g., severe dementia, epileptic encephalopathy).
* Acute neurological events in the perioperative period (e.g., stroke, intracranial hemorrhage).
* Severe hepatic dysfunction (Child-Pugh Class C).
* Participation in another interventional study potentially affecting sedation or cognitive outcomes.
* Pregnancy or lactation.
* Patients in whom short-term survival is deemed unlikely due to clinical course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to the ICU following cardiac surgery. These patients are expected to require invasive mechanical ventilation and continuous sedation for more than 6 hours postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of time spent in deep sedation | immediately after extubation or up to 48 hours of ICU sedation - whichever comes first
  BIS <50

SECONDARY OUTCOMES:
Duration of mechanical ventilation | immediately after extubation
Incidence of pulmonary infection | immediately after ICU discharge
  any kind of pulmonary infection, including tracheobronchitis, pneumonia
Incidence of ICU delirium | immediately after extubation
  assessed using CAM-ICU or ICDSC
Time average of vasopressor dose | immediately after extubation or after 48 hours of invasive ventilation
  Time average of Noradrenaline dose
ICU and hospital LOS | immediately after hospital discharge
  in days
in hospital mortality | immediately after hospital discharge
Incidence of BIS suppression events | immediately after extubation or after 48 hours of invasive ventilation
  episodes where the suppression ratio exceeds 10%, indicating potential over-sedation or EEG suppression

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Medical University Graz, Graz, Styria
  - Klinikum Wels, Wels, Upper Austria

IPD SHARING:
Plan to Share IPD: Undecided